CLINICAL TRIAL: NCT01094704
Title: Durability of Hypertonic Saline for Enhancing Mucociliary Clearance in Cystic Fibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Johns Hopkins University (Other); Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Scott Donaldson, MD, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 09-0670
Record Dates: First submitted 2010-03-19; First posted 2010-03-29 (Estimated); Results first posted 2012-08-21 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-08

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; mucociliary clearance; hypertonic saline
MeSH Terms: conditions — Cystic Fibrosis | interventions — Sodium Chloride; Saline Solution, Hypertonic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypertonic Saline - 1 hour (Experimental): sodium chloride (7%); mucociliary clearance measured 1 hour post dose
  Interventions: Drug: sodium chloride (7%)
- Hypertonic Saline - 4 hours (Experimental): sodium chloride (7%); mucociliary clearance measured four hours post-dose.
  Interventions: Drug: sodium chloride (7%)

INTERVENTIONS:
Drug: sodium chloride (7%) — 4mL nebulized 7% sodium chloride
  Other Names: Hyper-Sal; Hypertonic saline (7%)

SUMMARY:
Direct measurement of mucociliary and cough clearance (MCC/CC) has been used as a biomarker in cystic fibrosis (CF). Additional knowledge of the performance of this biomarker is needed to inform exploratory clinical trial design in support of programs to develop new inhaled therapies for CF. We hypothesize that MCC/CC measurements can be used to determine the durability of action of agents like hypertonic saline (HS) which increase epithelial lining fluid height.

DETAILED DESCRIPTION:
A reduction in epithelial lining fluid height in cystic fibrosis (CF) as a consequence of decreased function of the Cystic Fibrosis Transmembrane conductance Regulator (CFTR) chloride channel and related increased activity of the Epithelial sodium (Na) Channel (ENaC) results in impaired mucociliary clearance (MCC), mucus stasis, inflammation, infection, and ultimately progressive bronchiectasis. Inhalation of hypertonic saline (HS), through a direct osmotic effect on the airways, results in an increase in epithelial lining fluid height in vitro and an increase in MCC in vivo as measured following inhalation of a radiotracer with gamma scintigraphy (Sood, et al 2003). MCC as a biomarker is being validated in the clinic, as administration of inhaled hypertonic saline (HS) to cystic fibrosis patients results in short- and medium-term improvements in MCC (Donaldson, et al 2006), while long-term administration of HS is associated with improvements in the registration endpoints of lung function and pulmonary exacerbations (Elkins, et al 2006). Based in large part on these studies, HS has gained acceptance in the CF community, with estimates of up to 50% of patients being treated with this therapy. MCC/CC is thus an excellent choice as a Proof of Concept endpoint for exploratory clinical studies of ENaC modulators. Prior clinical experience with the ENaC blocker amiloride, which improves MCC acutely in healthy volunteers (Sood, et al 2003) but failed to improve lung function in long-term studies in CF (Pons, et al 2000), suggests that durable ENaC modulation will be required for clinical success. It is believed that modulation of ENaC for a period of at least 4 hours will be required to achieve the necessary durability. This durability should also enable twice daily dosing. For comparison we need to know the effectiveness of HS over this same period. Thus, this study is intended to assess 1) the duration of action out to 4 hours for inhaled hypertonic saline (7%) in adult CF patients and 2) the variability of MCC/CC measurements with and without HS treatment. These assessments at UNC will be compared to similar measures at Johns Hopkins University (JHU) for Novartis to determine the feasibility for future multicenter studies using MCC/CC as a primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Gender: Male or female (non-pregnant, non-lactating)
* Cystic fibrosis documented by a compatible clinical and radiographic presentation, and sweat chloride > 60 mEq/l or 2 disease causing CFTR mutations.
* Severity of Disease:

  1. Must have FEV1 of greater than or equal to 50% of predicted at the screening visit.
  2. Must have an oxygen saturation of >92% on room air as determined by pulse oximetry at the screening visit.
* Patient or legally authorized representative agrees to the patient/individual's participation in the study by signing and dating the informed consent form after the nature of the study has been fully explained and all questions have been satisfactorily answered.

Exclusion Criteria:

* Unstable lung disease: As defined by a change in medical regimen during the preceding 2 weeks; an FEV1 >15% below recent (within 6 months) clinical measurements; or a significant new finding on chest radiograph (pneumothorax, lobar/segmental collapse) not considered a part of the usual, chronic progression of CF lung disease.
* Patients unable or unwilling to be withdrawn from hypertonic saline therapy, dornase alfa, or N-acetylcysteine 3 days prior to and for the duration of each Baseline and Treatment Period will be excluded.
* Patients unable to withhold use of long-acting bronchodilators (i.e., Salmeterol, Advair, Formoterol), anti-cholinergics, and vest therapy 12 hours prior to and for the duration of each treatment period.
* Patients unable to withhold short-acting bronchodilator 6 hours prior to and for the duration of each treatment period except as prescribed by the study protocol.
* Patients that have received an investigational drug or therapy during the preceding 30 days.
* Patients that have had radiation exposure within the past year that would cause them to exceed Federal Regulations by participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Bennett, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina

REFERENCES:
- [Background] Donaldson SH, Bennett WD, Zeman KL, Knowles MR, Tarran R, Boucher RC. Mucus clearance and lung function in cystic fibrosis with hypertonic saline. N Engl J Med. 2006 Jan 19;354(3):241-50. doi: 10.1056/NEJMoa043891. PMID 16421365
- [Background] Elkins MR, Robinson M, Rose BR, Harbour C, Moriarty CP, Marks GB, Belousova EG, Xuan W, Bye PT; National Hypertonic Saline in Cystic Fibrosis (NHSCF) Study Group. A controlled trial of long-term inhaled hypertonic saline in patients with cystic fibrosis. N Engl J Med. 2006 Jan 19;354(3):229-40. doi: 10.1056/NEJMoa043900. PMID 16421364
- [Background] Bennett WD, Olivier KN, Zeman KL, Hohneker KW, Boucher RC, Knowles MR. Effect of uridine 5'-triphosphate plus amiloride on mucociliary clearance in adult cystic fibrosis. Am J Respir Crit Care Med. 1996 Jun;153(6 Pt 1):1796-801. doi: 10.1164/ajrccm.153.6.8665037.
- [Background] Donaldson SH, Boucher RC. Sodium channels and cystic fibrosis. Chest. 2007 Nov;132(5):1631-6. doi: 10.1378/chest.07-0288. PMID 17998363
- [Background] Pons G, Marchand MC, d'Athis P, Sauvage E, Foucard C, Chaumet-Riffaud P, Sautegeau A, Navarro J, Lenoir G. French multicenter randomized double-blind placebo-controlled trial on nebulized amiloride in cystic fibrosis patients. The Amiloride-AFLM Collaborative Study Group. Pediatr Pulmonol. 2000 Jul;30(1):25-31. doi: 10.1002/1099-0496(200007)30:13.0.co;2-c. PMID 10862159
- [Background] Sood N, Bennett WD, Zeman K, Brown J, Foy C, Boucher RC, Knowles MR. Increasing concentration of inhaled saline with or without amiloride: effect on mucociliary clearance in normal subjects. Am J Respir Crit Care Med. 2003 Jan 15;167(2):158-63. doi: 10.1164/rccm.200204-293OC. Epub 2002 Oct 31. PMID 12411282
- [Derived] Wark P, McDonald VM, Smith S. Nebulised hypertonic saline for cystic fibrosis. Cochrane Database Syst Rev. 2023 Jun 14;6(6):CD001506. doi: 10.1002/14651858.CD001506.pub5. PMID 37319354

RESULTS

PARTICIPANT FLOW:
Groups:
- Hypertonic Saline - 1 Hour: Single dose of hypertonic saline (7%) nebulized followed by MCC/CC assessment one hour post-dose.
- Hypertonic Saline - 4 Hours: Single dose of hypertonic saline (7%) nebulized followed by MCC/CC assessment four hours post-dose.
Period: Overall Study
Arm/Group | Hypertonic Saline - 1 Hour | Hypertonic Saline - 4 Hours
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hypertonic Saline - 1 Hour | Hypertonic Saline - 4 Hours | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Mucociliary Clearance (0-90 Minutes) at 1 and 4 Hrs Post Dose (MCC4hr - MCCbaseline; MCC1hr - MCCbaseline)
Description: Duration of action of hypertonic saline as determined by measurements of mucociliary clearance/cough clearance 4 hours post dose.
Time Frame: 1-4 hours post-dose
Population: ITT
Measure: Mean (Standard Deviation); unit: Absolute % change
Arm/Group | Hypertonic Saline - 1 Hour | Hypertonic Saline - 4 Hours
Number analyzed (Participants) | 8 | 8
Absolute % change | 5.9 (8.9) | 6.7 (14.4)

ADVERSE EVENTS:
Arm/Group | Hypertonic Saline - 1 Hour | Hypertonic Saline - 4 Hours
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less